CLINICAL TRIAL: NCT05311696
Title: Examining the Efficacy and Feasibility of a Residential Retreat Program for PTSD in First-responders and Veterans: A Non-randomized Controlled Study
Brief Title: Residential Retreat for Veterans and First-responders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Valhalla Project Niagara (Industry)
Responsible Party: Sponsor
Other Study IDs: 2650
Record Dates: First submitted 2022-03-03; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residential Cohort: Those completing the program in a residential context
  Interventions: Other: psychoeducation
- Online Cohort: Those completing the program online
  Interventions: Other: psychoeducation

INTERVENTIONS:
Other: psychoeducation — The program consists of psychoeducational material regarding PTSD, demonstration of various stress management techniques, and social cohesion activities
  Other Names: demonstration of stress management techniques; social cohesion activities

SUMMARY:
The purpose of this study is to determine the potential efficacy and feasibility of a residential retreat program to address PTSD symptoms in Veterans and First-responders

DETAILED DESCRIPTION:
After obtaining written consent, participants will complete their program as they had previously intended. Each wave of the residential retreat program will last 5 days. During the program, participants will complete the study questionnaires. They will complete these questionnaires again 1 month after the completion of the program. As a control, individuals completing the program in the online format will also be asked to provide written consent and will complete the questionnaires during the program and 1-month after its completion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD, being a military veteran or first-responder, awareness of treating physician about program attendance

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These are individuals who are veterans of the military of first-responders, who have also been diagnosed with PTSD.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-03-27 (Estimated); Primary Completion 2022-11-21 (Estimated); Study Completion 2023-11-21 (Estimated)

PRIMARY OUTCOMES:
Symptom Management of PTSD Using the Perceived Medical Condition Self-Management Scale | 1-month after completion of the program
  determining the potential efficacy of the residential program for improving symptom management. The scale is adapted to reflect participants management of their PTSD symptoms. Score ranges from 8 to 40. Higher scores indicate better management.
Drop-out rate in the Residential Program | at the end of the 5-day residential program for the residential cohort
  Determining the extent of treatment drop-out in the Residential Program
Symptoms of PTSD Indicated by the PTSD Checklist for DSM-5 scale. | 1-month after completion of the program
  determining the potential efficacy of the residential program for improving PTSD symptoms. Scores range from 0 to 80. Higher scores indicate more symptoms of PTSD.
Interpersonal and Intrapersonal Functioning Using the Brief Inventory of Psychosocial Functioning (B-IPF) | 1-month after the completion of the program
  determining the potential efficacy of the residential program for improving interpersonal and intrapersonal functioning (e.g., relationship with family, ability to manage daily tasks, etc.). Scores range from 0 to 42. Higher scores indicate more problems and lower functioning.
Drop-out rate in the Online Program | at the end of the 2 month online program for the online cohort.
  Determining the extent of treatment drop-out in the Online Program

CONTACTS AND LOCATIONS:
Overall Officials: Jaan Reitav, PhD, C.Psych, Principal Investigator — Canadian Memorial Chiropractic College
Locations (1):
- Valhalla Project Niagara, Niagara-on-the-Lake, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be available upon request by other researchers.